CLINICAL TRIAL: NCT03428646
Title: A Prospective Observational Study of Patients Receiving DUPIXENT® for Atopic Dermatitis
Brief Title: Study of Patients Receiving DUPIXENT® for Atopic Dermatitis (AD)
Acronym: PROSE
Status: Active, not recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: R668-AD-1762
Record Dates: First submitted 2017-12-13; First posted 2018-02-09 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Dermatitis, Atopic
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Biospecimen Retention: Samples With DNA — Optional sub-study: Blood samples will be collected and stored up to 10 years for future use in bio-marker research. Participants who agree to provide blood samples for future research will be required to sign a separate informed consent form (ICF) before collection of the samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dupilumab — Dupixent 1 dose at Baseline required for eligibility; otherwise, no therapeutic intervention required during the course of the study. In addition to (or substituting for) DUPIXENT®, participants may receive marketed drugs as deemed necessary by their physicians for the treatment of AD or comorbid conditions.
  Other Names: DUPIXENT®; REGN668

SUMMARY:
A long-term observational registry in patients with atopic dermatitis (AD) initiating treatment with DUPIXENT® (dupilumab)

DETAILED DESCRIPTION:
This is a prospective observational study conducted to (1) characterize the patients who receive DUPIXENT® for AD in a real world setting with respect to their medical history, socio-demographic and disease characteristics, and prior and concomitant treatments of AD; (2) characterize real world use patterns of DUPIXENT® for AD (eg, most commonly used regimens by line of therapy, reason for initiation of new treatments, concomitant therapies, treatment durations and reasons for discontinuation and/or switching); (3) assess the long-term effectiveness of DUPIXENT® in AD patients in a real world setting; (4) assess comorbid atopic conditions, patterns of use and effects of treatment in comorbid atopic conditions in patients who receive DUPIXENT® for AD; and (5) collect safety data on study participants

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, 12 years of age or older at the baseline visit. NOTE: Adolescent patients (at least 12 years old, but less than 18 years) are eligible in the US or Canada only after DUPIXENT receives the respective country's regulatory approval for use in this age group.
* Initiating treatment with DUPIXENT® as standard-of-care for AD according to the country-specific prescribing information (Note: Participants will be screened when they received their initial prescription for DUPIXENT®).
* Willing and able to comply with study-related activities.
* Able to understand and complete study-related questionnaires.
* Provide signed informed consent or parental/legal guardian consent plus patient assent, where applicable.

Key Exclusion Criteria:

* Patients who have a contraindication to the drug according to the country-specific prescribing information label.
* Any condition that, in the opinion of the investigator, may interfere with patient's ability to participate in the study, such as short life expectancy, substance abuse, severe cognitive impairment, or other co-morbidities that can predictably prevent the patient from adequately completing the schedule of visits and assessments.
* Prior use of dupilumab within 6 months of the screening visit, or within 6 months of the baseline visit if screening and baseline occur on the same day.

NOTE: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population comprises adult and adolescent patients (male or female, ≥12 years old), who are initiating treatment with DUPIXENT® for AD according to the country-specific prescribing information.
Sampling Method: Non-Probability Sample
Enrollment: 858 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Registry Assessment: Baseline Characteristics | At baseline (day when DUPIXENT treatment is initiated)
  Medical history
Registry Assessment: Baseline Characteristic | At baseline (day when DUPIXENT treatment is initiated)
  Socio-demographics

SECONDARY OUTCOMES:
Registry (Physician) Assessment: Body Surface Area Affected (BSA) by Atopic Dermatitis | Baseline to month 60
  Percentage of BSA affected by AD assessed for each major section of the body
Registry (Physician) Assessment: Eczema Area and Severity Index (EASI) | Baseline to month 60
  Measure used in clinical practice and clinical trials to assess the severity and extent of AD
Registry (Physician) Assessment: Overall Disease Severity scale | Baseline to month 60
  Questionnaire used to characterizing the severity of AD on a 4-point scale (0=No disease, 1=Minimal disease, 2=Mild disease, 3=Moderate disease, 4=Severe disease)
Registry (Participant) Assessment: Patient Oriented Eczema Measure | Baseline to month 60
  Questionnaire used in clinical practice and clinical trials to assess disease symptoms in children and adults
Registry (Participant) Assessment: Pruritus Numerical Rating Scales (NRS) | Baseline to month 60
  Individual NRS used to rate the intensity of pruritus using a 0 to 10 numeric rating scale.
Registry (Participant) Assessment: Skin Pain or Soreness NRS | Baseline to month 60
  Individual NRS used to rate skin pain and soreness using a 0 to 10 NRS
Registry (Participant) Assessment: Skin Feeling Hot NRS | Baseline to month 60
  Individual NRS used to rate the sensation of skin feeling hot (burning sensation) using a 0 to 10 NRS
Registry (Participant) Assessment: Skin Sensitivity NRS | Baseline to month 60
  Individual NRS used to rate skin sensitivity using a 0 to 10 NRS
Registry (Participant) Assessment: Sleep Disturbance NRS | Baseline to month 60
  Individual NRS used to report the severity of their sleep disturbance using a 0 to 10 NRS
Registry (Participant) Assessment: Global Assessment of Atopic Dermatitis scale | Baseline to month 60
  Rate of overall well-being on a 5-point scale.
Registry (Participant) Assessment: Dermatology Life Quality Index (DLQI) | Baseline to month 60
  Questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL) in adults
Registry (Participant) Assessment: Children's Dermatology Life Quality Index (CDLQI) | Baseline to month 60
  Questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on QOL in pediatrics.
Registry (Participant) Assessment: Work Productivity and Activity Impairment Questionnaire for AD (WPAI-AD) | Baseline to month 60
  Questionnaire to assess the impact of AD on productivity.
Registry (Participant) Assessment: Health Care Resource Utilization Questionnaire | Baseline to month 60
  Questionnaire regarding hospitalization, or emergency room/ urgent care center visits due to AD.
Registry (Participant) Assessment: Dermatitis Family Impact Questionnaire | Baseline to month 60
  Questionnaire to assess the impact of atopic eczema on the QOL of the parents and family members of affected children.
Registry (Participant) Assessment: Missed School Days | Baseline to month 60
  Questionnaire to assess the number of missed school days since the last study assessment of adolescent patients (aged ≥ 12 to < 18 years) who are enrolled in school.
Registry (Participant) Assessment: Juniper Asthma Control Questionnaire (ACQ-5) | Baseline to month 60
  5-question version of questionnaire to evaluate asthma control in registry patients with comorbid asthma.
Registry (Participant) Assessment: Allergic Rhinitis Visual Analog Scale (AR-VAS) | Baseline to month 60
  Questionnaire used as a validated measuring instrument for the documentation of symptoms and therapy monitoring in AR.
Registry (Participant) Assessment: Changes in Concurrent Conditions | Baseline to month 60
  Rate of change in any other condition(s) (other than eczema, asthma, and allergic symptoms) on a 2-point scale (Better or Worse).
Registry (Participant) Assessment: Overall Health State | Baseline to month 60
  Rate of overall state of health on a 5-point scale (Poor, Fair, Good, Very Good or Excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Regeneron Pharmaceuticals
Locations (92):
- United States (86):
  - Regeneron Investigational Site, Birmingham, Alabama
  - Regeneron Investigational Site, Gilbert, Arizona
  - Regeneron Investigational Site, Fountain Valley, California
  - Regeneron Investigational Site, Laguna Hills, California
  - Regeneron Investigational Site, Loma Linda, California
  - Regeneron Investigational Site, Los Angeles, California
  - Regeneron Investigational Site, Manhattan Beach, California
  - Regeneron Investigational Site, Newport Beach, California
  - Regeneron Investigational Site, Oceanside, California
  - Regeneron Investigational Site, Redondo Beach, California
  - Regeneron Investigational Site, Riverside, California
  - Regeneron Investigational Site, Roseville, California
  - Regeneron Investigational Site, San Diego, California
  - Regeneron Investigational Site, Santa Monica, California
  - Regeneron Investigational Site, Thousand Oaks, California
  - Regeneron Investigational Site, New Haven, Connecticut
  - Regeneron Investigational Site, Coral Gables, Florida
  - Regeneron Investigational Site, Margate, Florida
  - Regeneron Investigational Site, West Palm Beach, Florida
  - Regeneron Investigational Site, Atlanta, Georgia
  - Regeneron Investigational Site, Macon, Georgia
  - Regeneron Investigational Site, Marietta, Georgia
  - Regeneron Investigational Site, Sandy Springs, Georgia
  - Regeneron Investigational Site, Champaign, Illinois
  - Regeneron Investigational Site, Chicago, Illinois
  - Regeneron Investigational Site, La Grange Park, Illinois
  - Regeneron Investigational Site, Skokie, Illinois
  - Regeneron Investigational Site, Springfield, Illinois
  - Regeneron Investigational Site, Fort Wayne, Indiana
  - Regeneron Investigational Site, Plainfield, Indiana
  - Regeneron Investigational Site, Overland Park, Kansas
  - Regeneron Investigational Site, Corbin, Kentucky
  - Regeneron Investigational Site, Louisville, Kentucky
  - Regeneron Investigational Site, Rockville, Maryland
  - Regeneron Investigational Site, Towson, Maryland
  - Regeneron Investigational Site, Upper Marlboro, Maryland
  - Regeneron Investigational Site, White Marsh, Maryland
  - Regeneron Investigational Site, Quincy, Massachusetts
  - Regeneron Investigational Site, Ann Arbor, Michigan
  - Regeneron Investigational Site, Bay City, Michigan
  - Regeneron Investigational Site, Troy, Michigan
  - Regeneron Investigational Site, Warren, Michigan
  - Regeneron Investigational Site, Columbia, Missouri
  - Regeneron Investigational Site, Kirksville, Missouri
  - Regeneron Investigational Site, St Louis, Missouri
  - Regeneron Investigational Site, Lincoln, Nebraska
  - Regeneron Investigational Site, Henderson, Nevada
  - Regeneron Investigational Site, Las Vegas, Nevada
  - Regeneron Investigational Site, Brick, New Jersey
  - Regeneron Investigational Site, East Windsor, New Jersey
  - Regeneron Investigational Site, Edison, New Jersey
  - Regeneron Investigational Site, Piscataway, New Jersey
  - Regeneron Investigational Site, Elmhurst, New York
  - Regeneron Investigational Site, Forest Hills, New York
  - Regeneron Investigational Site, Garden City, New York
  - Regeneron Investigational Site, Kew Gardens, New York
  - Regeneron Investigational Site, Lake Success, New York
  - Regeneron Investigational Site, Manhasset, New York
  - Regeneron Investigational Site, Mineola, New York
  - Regeneron Investigational Site, Mount Vernon, New York
  - Regeneron Investigational Site, New York, New York
  - Regeneron Investigational Site, The Bronx, New York
  - Regeneron Investigational Site, Troy, New York
  - Regeneron Investigational Site, Concord, North Carolina
  - Regeneron Investigational Site, Akron, Ohio
  - Regeneron Investigational Site, Athens, Ohio
  - Regeneron Investigational Site, Bexley, Ohio
  - Regeneron Investigational Site, Marion, Ohio
  - Regeneron Investigational Site, Mason, Ohio
  - Regeneron Investigational Site, Tulsa, Oklahoma
  - Regeneron Investigational Site, Portland, Oregon
  - Regeneron Investigational Site, Blue Bell, Pennsylvania
  - Regeneron Investigational Site, Philadelphia, Pennsylvania
  - Regeneron Investigational Site, Sellersville, Pennsylvania
  - Regeneron Investigational Site, Yardley, Pennsylvania
  - Regeneron Investigational Site, Charleston, South Carolina
  - Regeneron Investigational Site, North Charleston, South Carolina
  - Regeneron Investigational Site, Bellaire, Texas
  - Regeneron Investigational Site, Dallas, Texas
  - Regeneron Investigational Site, Grapevine, Texas
  - Regeneron Investigational Site, San Antonio, Texas
  - Regeneron Investigational Site, Sugar Land, Texas
  - Regeneron Investigational Site, Arlington, Virginia
  - Regeneron Investigational Site, Norfolk, Virginia
  - Regeneron Investigational Site, Bellevue, Washington
  - Regeneron Investigational Site, Milwaukee, Wisconsin
- Canada (6):
  - Regeneron Investigational Site, Hamilton, Ontario
  - Regeneron Investigational Site, Markham, Ontario
  - Regeneron Investigational Site, Ottawa, Ontario
  - Regeneron Investigational Site, Peterborough, Ontario
  - Regeneron Investigational Site, Toronto, Ontario
  - Regeneron Investigational Site, Québec

REFERENCES:
- [Derived] Bhatia N, Lynde CW, Fonacier L, Shao L, Bosman K, Korotzer A. Complete/Near-Complete Itch Response Observed in Patients with Moderate-to-Severe Atopic Dermatitis Initiating Dupilumab: 3-Year, Real-World, Interim Data from the PROSE Registry. Dermatol Ther (Heidelb). 2025 Jun;15(6):1523-1531. doi: 10.1007/s13555-025-01395-1. Epub 2025 Apr 15. PMID 40234297
- [Derived] Simpson EL, Lockshin B, Lee LW, Chen Z, Daoud M, Korotzer A. Real-World Effectiveness of Dupilumab in Adult and Adolescent Patients with Atopic Dermatitis: 2-Year Interim Data from the PROSE Registry. Dermatol Ther (Heidelb). 2024 Jan;14(1):261-270. doi: 10.1007/s13555-023-01061-4. Epub 2024 Jan 4. PMID 38175364
- [Derived] Bagel J, Nguyen TQ, Lima H, Jain N, Pariser DM, Hsu S, Yosipovitch G, Zhang H, Chao J, Bansal S, Chen Z, Richman D, Korotzer A, Ardeleanu M. Baseline Demographics and Severity and Burden of Atopic Dermatitis in Adult Patients Initiating Dupilumab Treatment in a Real-World Registry (PROSE). Dermatol Ther (Heidelb). 2022 Jun;12(6):1417-1430. doi: 10.1007/s13555-022-00742-w. Epub 2022 May 20. PMID 35590038